CLINICAL TRIAL: NCT00757718
Title: Sleep Disordered Breathing and Gestational Hypertension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Saskatchewan (Other)
Responsible Party: John K. Reid, Assistant Professor of Medicine, University of Saskatchewan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Bio: 08-21
Record Dates: First submitted 2008-09-22; First posted 2008-09-23 (Estimated); Last update posted 2009-09-09 (Estimated); Status verified 2009-09

CONDITIONS: Sleep Disordered Breathing; Obstructive Sleep Apnea; Gestational Hypertension; Preeclampsia
Keywords: Sleep Disordered Breathing; Obstructive Sleep Apnea; Gestational Hypertension; Preeclampsia
MeSH Terms: conditions — Sleep Apnea Syndromes; Sleep Apnea, Obstructive; Hypertension, Pregnancy-Induced; Pre-Eclampsia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- CPAP treatment (Active Comparator): Subjects will have repeat polysomnography on the second night, while wearing a continuous positive airway pressure (CPAP) device. Morning bloodwork will be drawn for inflammatory mediators.
  Interventions: Device: CPAP
- Oral appliance (Experimental): Subjects will have repeat polysomnography on the second night, while wearing an oral appliance, as well as a Breathe-Right nasal strip. Morning bloodwork will be drawn for inflammatory mediators.
  Interventions: Device: Oral Appliance

INTERVENTIONS:
Device: CPAP — One half of the subjects will be randomly assigned to wear continuous a positive airway pressure device on the second night of the study. Portable polysomnography will be repeated for this night and morning bloodwork for inflammatory markers will be repeated.
  Other Names: Respironics M Series Autoset CPAP; Somnoguard AP oral apliance; Breathe Right Nasal Srip
  Arms: CPAP treatment
Device: Oral Appliance — Half of the subjects will be assigned to wear an oral appliance and nasal strip on the second night of the study. Repeat portable polysomnography will be performed and morning bloodwork will again be drawn for inflammatory markers.
  Other Names: Somnoguard AP; Breathe Right nasal strip
  Arms: Oral appliance

SUMMARY:
Sleep disordered breathing (SDB) is a common problem in the adult population. By conservative estimates, 4% of the adult female population has SDB. SDB is a recognized cause of hypertension and treating SDB can improve blood pressure control in people with hypertension. More recently, research efforts have looked at SDB as a possible cause of pregnancy induced hypertension (PIH), a condition which complicates 10% of pregnancies. Traditionally, the best way to assess SDB required patients to spend a night sleeping in the Sleep Laboratory. This is inconvenient and for pregnant women often impossible to arrange, considering the short time frame that exists between time of PIH diagnosis and eventual delivery. Researchers at the University of Saskatchewan are now looking at whether an adequate sleep assessment can be performed at the bedside - either in a patient's home or on the hospital ward. The researchers will also look at different treatment options for sleep apnea, to see if these can improve blood pressure control in this patient population, and delay the need for early delivery. The information from this study may result in a detailed sleep assessment becoming part of the complete assessment of women with PIH. There is an association between sleep disordered breathing (SDB) and gestational hypertension (GHTN). Treatment for the SDB may represent an effective addition to the management of the cardiovascular and metabolic perturbations of GHTN We plan to assess women whether treating SDB with one of two methods will improve the management of GHTN. We will also assess if one method is more effective than the other.

ELIGIBILITY:
Inclusion Criteria:

* Women with singleton pregnancies who have the diagnosis of gestational hypertension.

Exclusion Criteria:

* Inability to comply with study parameters
* Delivery expected within 48 hours

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 26 (Estimated)
Dates: Start 2008-12; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Effectiveness of the two treatment arms at treating sleep disordered breathing. | single night

SECONDARY OUTCOMES:
Effectiveness of the treatment arms at improving metabolic perturbations of GHTN. | single night
Acceptability of therapy | single night

CONTACTS AND LOCATIONS:
Overall Officials: John K Reid, MD, Principal Investigator — University of Saskatchewan
Locations (1):
- Royal University Hospital, Saskatoon, Saskatchewan, Canada